CLINICAL TRIAL: NCT06059872
Title: What Makes a Responder, a Responder? Biomarkers to Help Identify Responders and Resistors to High-intensity Interval Training for Lower Extremity Chronic Stroke
Brief Title: Biomarkers of Reaction To HIIT Exercise
Acronym: BReaTHE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N4537-R; I01RX004537 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Stroke Rehabilitation; Lower Extremity Weakness, Spastic; Walking, Difficulty
Keywords: Predictors of Stroke Rehabilitation; Biomarkers of Stroke Rehabilitation; Exercise Intervention; Neuroimaging
MeSH Terms: conditions — Stroke; Paraparesis, Spastic; Mobility Limitation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: The investigators will enroll 55 Veterans with chronic subcortical stroke in the 12-week HIIT intervention, with the expectation that 48 participants (85%) will complete the entire program. In our experience, 65% of participants will respond to the HIIT intervention, resulting in an estimated 31 responders and 17 resistors. Each chronic subcortical stroke participant will be asked to participate in the overall study protocol with pre-, during-, and post-intervention measurements. The HIIT consists of three weekly 25-60 minute cycling sessions for 12 weeks at the Atlanta VA, administered by a trained exercise physiologist, for a total of 36 HIIT sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic Stroke with lower limb disability (Experimental): The investigators will enroll 55 Veterans with chronic subcortical stroke in the 12-week HIIT intervention, with the expectation that 48 participants (85%) will complete the entire program. In our experience, 65% of participants will respond to the HIIT intervention, resulting in an estimated 31 responders and 17 resistors. Each chronic subcortical stroke participant will be asked to participate in the HIIT study protocol. Classification of resistor or responder: A responder to the 12-week HIIT intervention will be defined as a participant who increases their walking speed to greater than 0.6 m/s. A resistor to the intervention will be defined as a participant who does not increase their walking speed to greater than 0.6 m/s.
  Interventions: Other: High Intensity Interval Training (HIIT)

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) — HIIT consists of three weekly 25-60 minute cycling sessions for 12 weeks at the Atlanta VA, administered by a trained exercise physiologist, for a total of 36 HIIT sessions.

SUMMARY:
Stroke survivors with lower limb disability can improve their walking speed with high-intensity interval training (HIIT) rehabilitation therapy. However, some individuals may not respond to HIIT even when fully adherent to the program. To address this, the investigators propose to build a predictive model that identifies if a Veteran with chronic subcortical stroke will improve their walking speed with HIIT by incorporating blood lactate as an early predictor of exercise response, and inhibitory neurotransmitter gamma-aminobutyric acid (GABA) and regional cerebral blood flow (CBF) as predictors of the brain's potential to respond, while also taking into consideration other factors such as comorbidities, demographics, and fitness levels.

DETAILED DESCRIPTION:
Most chronic subcortical stroke survivors have difficulty walking, but few predictors can help identify if a patient will respond to an exercise regimen and improve their function. To enhance precision rehabilitation for chronic subcortical stroke patients, personalized aerobic exercise interventions are crucial. This requires the development of innovative technologies that can identify the essential neurobiological factors to predict intervention response and enable clinicians to determine individualized rehabilitation targets. Lactate is one exciting new target that acts as a molecular messenger between the periphery and the brain. For lactate to have an impact on other organs, including the brain, there must be a substantial increase in its level in the bloodstream from baseline. When the blood lactate threshold is surpassed during exercise, lactate acts on the brain metabolically via the TCA cycle. Embedded within the TCA cycle is the means to increase or decrease neurotransmitter concentrations such as GABA and glutamate. Gamma-aminobutyric acid (GABA), the brain's major inhibitory neurotransmitter, is a new treatment target that promotes neural plasticity during stroke rehabilitation. Drawing from the framework of personalized rehabilitation approaches and our preliminary data, the investigators propose to build a predictive model that can identify if a chronic subcortical stroke patient will respond to exercise training. This model aims to predict improvements in walking speed by incorporating blood lactate as an early predictor of exercise response and GABA and cerebral blood flow (CBF) as predictors of the brain's potential to respond, in addition to other influencing factors such as comorbidities, demographics, and fitness levels. The overarching hypothesis is that robust neurophysiological factors driven by lactate can differentiate responders from resistors and that these factors can be applied clinically as biomarkers to predict functional outcomes after a 12-week HIIT intervention. The investigators will assess improvements in walking speed in 48 Veterans with lower limb disability due to chronic subcortical stroke in response to a 36-session (12-week) HIIT intervention. After the intervention, each adherent participant who improves their walking speed to greater than 0.6 m/s will be categorized as a responder while each adherent participant who does not improve their walking speed will be categorized as a resistor. At baseline and after 12 weeks of HIIT the investigators will evaluate walking speed, balance, leg strength, and endurance to identify resistors and responders to HIIT and collect a) GABA from the primary sensory-motor leg area using single-voxel magnetic resonance spectroscopy, b) CBF from the whole brain using pseudo-Continuous Arterial Spin Labeling MRI and c) VO2 max to evaluate change in CRF. During the intervention, the investigators will collect blood lactate via finger prick during sessions 1, 4, 7, 10, and 28 to assess its potential as an early predictor of exercise response. In aim 1 the investigators determine if surpassing the lactate threshold during the first 4 weeks of HIIT predicts the change in walking speed to 0.6 m/s, from pre- to post-HIIT. If lactate proves to be a robust early marker of functional response to exercise, the investigators will have an easy-to-deploy predictor of who will best benefit from HIIT. In aim 2 the investigators will determine if (a) baseline GABA and/or CBF predict improvements in walking speed from baseline to after HIIT and (b) if a change in GABA and/or CBF relate to a change in walking speed. The investigators aim to establish neurophysiological correlates of improving function with HIIT to better understand the mechanisms. Finally, in aim 3 the investigators will a predictive machine learning algorithm of who will improve their walking speed with HIIT using factors of blood lactate, baseline GABA and CBF, baseline leg weakness and VO2-max, pre-stroke fitness, age, sex, and comorbidities. The overarching objective is to develop a model to predict which Veteran with chronic stroke will respond to a 12-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

* chronic left or right subcortical stroke as defined by 6 months or more after a cardiovascular accident
* lower extremity motor impairment due to stroke that causes a walking speed of less than 0.6 m/s during a 10m walk
* Veteran status

Exclusion Criteria:

* MRI contraindications, including implanted cardiac pacemakers and severe claustrophobia
* any neurodegenerative condition other than stroke that may lead to lower extremity impairment
* a visual or auditory impairment that may hinder study procedures
* any medical condition that would preclude participation in a physical exercise intervention program

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
10 m walk test on a GAITRite mat | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To assess short-distance walking speed and gait characteristics.
Timed-Up-and-Go (TUG) test | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To assess short-distance walking and postural control.
6-minute walk test | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To assess endurance.

SECONDARY OUTCOMES:
Blood lactate change during HIIT session | On exercise day 1, 4, 7, 10, and 28. The total number of exercise days is 36 (3 times per week for 12 weeks).
  To assess if the participant increases their blood lactate during the HIIT session.
MEGA-PRESS Magnetic Resonance Spectroscopy | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To assess GABA from the ipsilesional and contralesional leg areas of the brain.
pseudo Continuous Arterial Spin Labeling MRI | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To assess whole brain regional cerebral blood flow.
Graded treadmill or bike testing | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To estimate VO2-max.

OTHER OUTCOMES:
Repetition max strength test | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To assess the leg strength of the affected and less affected leg.
Global physical activity questionnaire (GPAQ) | baseline (week 1)
  To assess pre-stroke fitness levels.
Self-administered Comorbidity Questionnaire (SCQ) | baseline (week 1) and after the completion of 12 weeks of exercise (week 14)
  To assess the presence and burden of comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Krishnamurthy, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Per VA guidelines and regulations, deidentified data will be shared upon written request to the PI.
Supporting Information: Study Protocol, ICF
Time Frame: Upon close of the study.